CLINICAL TRIAL: NCT00724074
Title: The Use of Continuous Wound Infusion Analgesia in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Health, Canada (Other)
Responsible Party: Dr. Gordon Arnett, Capital Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: garnett
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Total Knee Arthroplasty
Keywords: Arthritis of the knee; Knee replacement; Osteoarthritis, knee; Arthroplasty, knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S (Experimental): Patients receive the On-Q local continuous wound infusion system intra-operatively and use it for up to three days post-operatively.
  Interventions: Device: On-Q PainBuster with Bupivacaine
- C (Active Comparator): Usual care - post operative pain medications as per the knee arthroplasty care map.
  Interventions: Device: Usual Care

INTERVENTIONS:
Device: On-Q PainBuster with Bupivacaine — On-Q PainBuster continuous wound infusion analgesia system, using bupivacaine as the local anaesthetic
  Arms: S
Device: Usual Care — Usual Care
  Arms: C

SUMMARY:
The main purpose of this study is to determine if there is improvement in pain and other patient outcomes when using a continuous wound analgesia system after total knee replacement, compared to usual methods of pain control. Another purpose is to determine if the system makes it easier for nurses to care for these patients.

DETAILED DESCRIPTION:
Continuous local wound infusion analgesia is a relatively new way of managing post-operative pain, whereby a local anesthetic is continuously infused into the surgical area. Some studies and users have reported decreased pain, decreased opioid use, decreased post-operative nausea and vomiting, decreased length of stay, and improved patient and caregiver satisfaction with the use of continuous local wound infusion analgesia, when compared to placebo, or usual care, in arthroplasty and other surgical interventions.

Hypotheses:

Primary:

The On-Q PainBuster (continuous wound infusion analgesia) in TKA will result in improved patient pain control, compared to usual care.

Secondary:

* Pain scores post-operatively will be better than usual care.
* Fewer narcotics will be ingested post-operatively than with usual care.
* Post-op nausea and vomiting will be less than usual care.
* Length of stay will be shorter compared to usual care.
* Patient satisfaction will be greater than satisfaction with usual care.
* Post-operative infection rates will be no different between groups.
* Fall rates will be no different between groups.
* Subjects will participate in physical therapy the day of surgery.
* Nursing Intensity requirements will be less with the wound infusion due to fewer requests for pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for TKA at the Royal Alexandra Hospital
* Patient of Dr. Arnett
* Deemed fit for continuous wound infusion (no allergies to Bupivacaine or related medications) by anesthesia
* Cognitively aware, and provides informed consent
* Elective (not trauma-related) surgery
* Able to read, speak and understand English
* Adult < 70 years of age
* Intra-operative spinal anaesthesia
* Reside within metropolitan Edmonton, in a bungalow
* Have a caregiver at home
* ASA risk classification of 1 or 2
* Do not regularly use opioid medication pre-operatively
* Have preoperative knee range of motion > 90 degrees
* Body Mass Index < 40
* No known hepatic or liver insufficiency

Exclusion Criteria:

* Deemed unfit for continuous wound infusion due to allergies
* Other exclusion criteria to be determined

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Pain, measured by the 11-point numerical pain rating scale | Post-operatively for three days then again at follow-up

SECONDARY OUTCOMES:
Post-operative nausea and vomiting | Post-operatively for three days
Narcotic medications taken | Post-operatively for three days
Time to first mobilization, first transfer and first 30-M walk | Up to three days post-operatively
Number of adverse events | Three days post-op (observed) then at follow-up (self-report)
Length of Stay | Time of surgery to discharge
Satisfaction (patient and caregiver) | Discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Arnett, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada